CLINICAL TRIAL: NCT01825395
Title: Use of 3,4-Diaminopyridine(3 4-DAP)in the Treatment of Lambert-Eaton Syndrome (LEMS)
Brief Title: Use of 3,4-Diaminopyridine in the Treatment of Lambert-Eaton Syndrome
Acronym: 3 4-DAP
Status: Approved for marketing | Type: Expanded Access
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 04-0567
Record Dates: First submitted 2013-03-22; First posted 2013-04-05 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Lambert Eaton Myasthenic Syndrome
MeSH Terms: conditions — Lambert-Eaton Myasthenic Syndrome

INTERVENTIONS:
Drug: 3, 4-Diaminopyridine

SUMMARY:
To learn more about the effect of 3, 4-Diaminopyridine (3,4-DAP) on patient diagnosed with Lambert-Eaton myasthenic syndrome (LEMS).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older,
* Diagnosed with LEMS,
* If female, have a negative pregnancy test, and
* If premenopausal, be willing to practice an effective form of birth control during the study,
* Tested and found by ECG not to have a prolonged QT syndrome,
* Agree to have a second ECG at the time of peak drug effect,
* Has understood and signed the Informed Consent.

Exclusion Criteria:

* Is known to have a sensitivity to 3, 4-DAP,
* Has a history of:

  1. past or current seizures,
  2. cardiac arrhythmia,
  3. hepatic, renal or hematologic disease, or
  4. severe asthma,
* Is believed by the investigator to be unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Steven P Ringel, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States